CLINICAL TRIAL: NCT03566680
Title: Treating Contact Lens Discomfort With Orthokeratology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OAN 000520524
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Results first posted 2020-05-05 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Dry Eye; Contact Lens Complication
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All subjects will be fit in orthokeratology contact lenses and be monitored for three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Orthokeratology Group (Experimental): All subjects will be fit in orthokeratology contact lenses.
  Interventions: Device: Orthokeratology

INTERVENTIONS:
Device: Orthokeratology — Orthokeratology is a type of contact lens that is worn over night to reduce refractive error, so patients do not need to wear vision correction during the day.

SUMMARY:
The primary aim of this study is to understand if orthokeratology can be used to improve contact lens comfort and the secondary aim is understand patient adaptation to orthokeratology.

DETAILED DESCRIPTION:
Orthokeratology has yet to be fully explored for the treatment of contact lens discomfort (CLD), though some support for this practice exists in the literature. Carracedo et al., Lipson et al., and Garcia-Porta et al. found that orthokeratology resulted in better ocular comfort than soft contact lenses. Nevertheless, all three studies excluded subjects who had been diagnosed with dry eye and all three studies used symptoms surveys that were not specific to assessing CLD. Garcia-Porta et al.'s study was also limited by including both neophytes and established contact lens wearers. Yet, these studies overall suggest that orthokeratology could be used as a treatment for CLD, and one case report has even found that orthokeratology is a viable option for treating contact lens intolerance.

To date, there has yet to be a study fully investigating orthokeratology as an alternative to soft contact lens use in patients with CLD. Therefore, the purpose of this study is to formally investigate if orthokeratology is a good alternative to soft contact lenses for patients who are experiencing CLD or for patients who have dropped out of contact lenses because of CLD. This study will also simultaneously evaluate the neophyte orthokeratology wearing experience with hopes of finding additional means for improving contact lens comfort. Knowing the success of orthokeratology in wearers with CLD will allow practitioners to better help and prescribe for those who may have experienced or at risk for experiencing CLD. It may also be a way to allow patients additional years of contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

* A completed comprehensive eye exam within the past two years
* Contact lens discomfort or discontinuation of contact lenses because of discomfort within the past 6 months
* Able to wear the Emerald™ Contact Lens (Oprifocon A, Euclid Systems Corporation)
* Refractive error better than -5.00 diopters with less than 1.50 diopters of cylinder
* Keratometry values between 40.00 D and 46.00 D

Exclusion Criteria:

* Past orthokeratology use
* Ocular surgery within the past 12 months
* History of severe ocular trauma
* Active ocular infection or inflammation
* Ocular disease other than dry eye
* Accutane or ocular medication use
* Pregnant or breast feeding
* A condition or situation that may put the subject at significant risk, confound the study results, or may significantly interfere with study participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pucker, OD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
The data will be shared in aggregate as a published manuscript.

REFERENCES:
- [Derived] Duong K, McGwin G Jr, Franklin QX, Cox J, Pucker AD. Treating Uncomfortable Contact Lens Wear With Orthokeratology. Eye Contact Lens. 2021 Feb 1;47(2):74-80. doi: 10.1097/ICL.0000000000000690. PMID 32097182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited if they were in the 18-45 had significant Contact lens dry eye questionnaire 8 (cldeq-8) scores (12 or greater), subjects also had to be previous spectacle or contact lens wearers, and had relatively healthy meidcal history, as well as being able to be fit within the approved fda range for orthok (orthokeratology) lenses.
Groups:
- Orthokeratology Group: All subjects will be fit in orthokeratology contact lenses.
  Orthokeratology: Orthokeratology lenses are a type of lens that can be worn overnight while a patient is sleeping, during this time the cornea is reshaped by the lens thus reducing the refractive error. This allows subjects to have corrected vision during the day, this would prevent the need of wearing contact lenses or glasses throughout the course of the day.
Period: Overall Study
Arm/Group | Orthokeratology Group
Started | 46
Completed | 29
Not Completed | 17
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All subjects who fit the screening criteria 18-45 years old, with adequate cldeq-8 scores, and good overall health were allowed to participate in this study regardless of sex race or ethnicity.
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: Years] | 24.22 [18 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Comfort
Description: Contact lens comfort was measured with the Contact Lens Dry Eye Questionnaire-8 (Range = 0 to 28 with lower scores being better). Subjects were required to have Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) scores of 12 or greater in order to participate in this study.
Time Frame: 1 Month Compared to Baseline
Population: Participants recruited for this study were required to be within the age ranges of 18-45 with good overall health. Subjects were required to need vision correction, and willing to come in for multiple in person visits during the first month of enrollment.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
Units on a Scale
  Baseline | 22.03 (5.47)
  1 Month | 9.83 (5.37)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Contact Lens Comfort
Description: Contact lens comfort was measured with the Contact Lens Dry Eye Questionnaire-4 (Range = 0 to 18 with lower scores being better).
Time Frame: 1 Week Compared to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
score on a scale
  Baseline | 11.72 (2.59)
  1 week | 7.44 (3.55)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Contact Lens Comfort
Description: Eye comfort will be measured with the Contact Lens Dry Eye Questionnaire-4 (Range = 0 to 18 with lower scores being better).
Time Frame: 3 Month Compared to Baseline
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
Score on a Scale
  Baseline | 11.72 (2.59)
  3 months | 4.27 (3.52)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Non-Invasive Tear Break-Up Time
Description: This is a measure of tear stability (Measured in seconds with higher amounts of time being better).
Time Frame: 1 Month Compared to Baseline
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
Seconds
  Baseline | 12.25 (6.28)
  1 month | 12.60 (5.67)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p = 0.73, t-test, 2 sided

5. Secondary Outcome: Tear Meniscus Height
Description: This is a measure of tear volume (Measured in millimeters with higher heights being better).
Time Frame: 1 Month Compared to Baseline
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
Millimeters
  Baseline | 0.27 (0.09)
  1 Month | 0.26 (0.07)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p = 0.08, t-test, 2 sided

6. Secondary Outcome: Phenol Red Thread
Description: This is a measure of tear volume (Range = 0 to 75 millimeters with higher values being better).
Time Frame: 1 Month Compared to Baseline
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Orthokeratology Group
Number analyzed (Participants) | 29
Millimeters
  Baseline | 25.75 (9.19)
  1 Month | 27.67 (8.57)
Statistical Analysis 1: Comparison: Orthokeratology Group; Test type: Equivalence; p = 0.72, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects were required to come in for four in person visits over the course of the first month of this study. However an email containing a survey was sent out after 3 months prior to the subject being exited from the study. During this time subjects were encouraged to contact the Pucker laboratory directly regarding any issues or questions they had about their orthok lenses or their general vision.
Arm/Group | Orthokeratology Group
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03566680/Prot_SAP_ICF_000.pdf